CLINICAL TRIAL: NCT05352867
Title: Phase Ⅱ Clinical Trial to Evaluate the Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (LVRNA009) in Chinese People Aged 18~59 Years
Brief Title: Clinical Trial of SARS-CoV-2 mRNA Vaccine in Chinese People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LVRNA009-Ⅱ-01
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — LVRNA009 COVID-19 vaccine; Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50μg group (Experimental)
  Interventions: Biological: SARS-CoV-2 (LVRNA009) 50μg group
- 100μg group (Experimental)
  Interventions: Biological: SARS-CoV-2 (LVRNA009) 100μg group
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 (LVRNA009) 50μg group — 50μg/person
  Arms: 50μg group
Biological: SARS-CoV-2 (LVRNA009) 100μg group — 100μg/person
  Arms: 100μg group
Other: Placebo — 0.5ml/person
  Arms: Placebo

SUMMARY:
Phase Ⅱ Clinical Trial to Evaluate the Safety and Immunogenicity of the New Coronavirus mRNA Vaccine (LVRNA009) in Chinese People Aged 18~59 Years

ELIGIBILITY:
Inclusion Criteria:

1. The age at the time of the first dose of the vaccine is 18-59 years old, and the gender is not limited;
2. The subject has full capacity for civil conduct;
3. Axillary body temperature is less than 37.3 ℃ on the day of enrollment;
4. Subjects have independent judgment ability, can read, understand and complete vaccination diary cards, and they participate voluntarily and sign an informed consent form.

Exclusion Criteria:

1. The subject has a history of contact with a person infected with SARS-CoV-2 (positive nucleic acid test) or a person suspected of being infected within 14 days;
2. Have a history of severe allergies to any vaccines, foods, and drugs, such as urticaria, anaphylactic shock, skin eczema, allergic dyspnea, angioedema, etc.;
3. The subject has a history of hypersensitivity to any component of the study vaccine (SARS-CoV-2 mRNA, Dlin-MC3-DMA, cholesterol, distearoylphosphatidylcholine, PEG2000-DMG, phosphate buffer);
4. Have a history of SARS virus infection;
5. Those with a medical history or family history of epileptic convulsions or convulsions, neurological diseases and mental diseases;
6. There is a history of thrombocytopenia or other coagulation disorders diagnosed by the hospital before enrollment;
7. The investigator judges that they are known or suspected to suffer from more serious diseases at the same time, including: respiratory diseases, tuberculosis, acute infection or active chronic disease, liver and kidney disease, cardiovascular disease (cardiopulmonary failure), and drug-uncontrollable hypertension (systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg), malignant tumor, infection or allergic skin disease, HIV infection (test report can be provided);
8. Congenital malformations, developmental disorders, or chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders, Guillain-Barré syndrome) determined by the investigator to be unsuitable for participating in this research;
9. Those with known immunological impairment or low function diagnosed by the hospital before enrollment;
10. There is evidence that he is a smoker, alcohol abuser and drug abuser;
11. Positive SARS-CoV-2 nucleic acid test results and/or positive antibody test results before the first dose of vaccination;
12. Female: a person with a positive urine pregnancy test, who is pregnant, breastfeeding, or has a pregnancy plan within 1 year; male: a person whose spouse has a pregnancy plan within 1 year;
13. Any other investigational or unregistered product (drug, biological product, or device) is being used before the first dose of vaccine, or is planned to be used during the study;
14. Those who received immune enhancement or immunosuppressive therapy within 6 months before the first dose of vaccine (continuous oral or infusion for more than 14 days);
15. Has been diagnosed with congenital or acquired immunodeficiency, or suspected of having a systemic disease that may interfere with the conduct or completion of the study, such as: tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV); ), syphilis infection, etc.;
16. Those who have received whole blood, plasma and immune globulin treatment within 6 months before the first dose of vaccine;
17. Received other inactivated vaccines within 14 days before the first dose of vaccine, and received live attenuated vaccines within 28 days;
18. Antipyretic, analgesic and anti-allergic drugs are being used within 3 days before enrollment;
19. Subjects who, in the judgment of the investigator, cannot follow the research procedures, abide by the agreement, or plan to permanently relocate from the local area before the end of the study, or plan to leave the local area for a long time during the scheduled visit;
20. The relevant staff members involved in this research or their immediate family members (such as spouses, parents, siblings or children);
21. According to the judgment of the investigator, there are other circumstances that are not suitable for participating in this clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Level of SARS-CoV-2 novel coronavirus S protein antibody (IgG) | 28 days after full-vaccination
Level of SARS-CoV-2 novel coronavirus neutralizing antibodies | 28 days after full-vaccination

SECONDARY OUTCOMES:
Incidence of adverse events | 14 days and 28 days after each dose of vaccination
Incidence of adverse events associated with the experimental vaccine | 14 days and 28 days after each dose of vaccination
Incidence of SAEs | 28 days, 3 months, 6 months and 12 months after first vaccination to full vaccination
Incidence of SAEs associated with the experimental vaccine | 28 days, 3 months, 6 months and 12 months after first vaccination to full vaccination
Incidence of grade ≥3 adverse events | 28 days after each dose or full vaccination
Incidence of grade ≥3 adverse events associated with the experimental vaccine | 28 days after each dose or full vaccination
Withdrawal from the trial due to adverse events | 28 days after each dose or full vaccination
Level of SARS-CoV-2 novel coronavirus S protein antibody (IgG) | 14 days, 3 months, 6 months and 12 months after full vaccination
Positive conversion rate of SARS-CoV-2 novel coronavirus S protein antibody | 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Level of SARS-CoV-2 novel coronavirus neutralizing antibody | 14 days, 3 months, 6 months and 12 months after full vaccination
Positive conversion rate of SARS-CoV-2 novel coronavirus neutralizing antibody | 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Level of specific cellular immune response against the new coronavirus (2019-nCoV) in subjects participating in cellular immune blood collection（IL-2、IL-4、IL-13、IFN-γ ）（ELISPOT） | 7th day after full vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Outpatient Department of Hunan Provincial Center For Disease Control And Prevention, Changsha, Hunan
  - Xiangtan Center For Disease Control And Prevention, Xiangtan, Hunan